CLINICAL TRIAL: NCT02530944
Title: Web-based Genetic Research on Lupus
Status: Completed | Type: Observational
Sponsor: 23andMe, Inc. (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 23andMe_SLE001
Record Dates: First submitted 2015-08-18; First posted 2015-08-21 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Lupus; Systemic Lupus Erythematosus (SLE); genetic; online; genome wide association; systemic lupus erythematosus; genome wide association study (GWAS)
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples are collected for DNA analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lupus patients: People diagnosed with Systemic Lupus Erythematosus by a physician

SUMMARY:
The goal of this new lupus research study is two-fold: first, to understand the genetic associations found between people's DNA and this disease, and second, to apply this understanding to drug development efforts with the investigator's partners at Pfizer.

DETAILED DESCRIPTION:
Lupus is a difficult disease to diagnose and one that's difficult to manage, given the lack of specific medicines to treat lupus and the side-effects of current medications. The investigators believe genetics may play a critical role in developing better lupus diagnoses and treatments. If individuals are eligible to participate, the investigators will send a 23andMe DNA saliva kit at no cost. Participants will be asked to take a 15 minute online survey with questions about their lupus experience, symptoms and response to treatments, in addition to five additional bi-monthly short surveys and one final study survey during the 12-month participation. Learn more and join the lupus study today: https://www.23andme.com/lupus/

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with lupus by a qualified physician.
* consents to have 23andMe (via a partner) contact the physician to obtain medical record information
* willing to submit a saliva sample for DNA testing and complete online surveys related to condition
* at least 6 years old (minors under 18 require parental consent to enroll)
* access to the internet
* resides in the United States

Exclusion Criteria:

-

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2015-05; Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Salivary DNA sample for genetic analysis | 12 months
Online survey | 12 months
  Questions about lupus experience, symptoms and response to treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Www.23Andme.Com/Lupus, Mountain View, California, United States